CLINICAL TRIAL: NCT00443729
Title: A Multicenter, Double-Blind, Randomized, Active-Controlled Study to Evaluate the Safety and Antiretroviral Activity of MK0518 Versus KALETRA in HIV-Infected Patients Switched From a Stable KALETRA-Based Regimen - Study B
Brief Title: MK0518 in the Treatment of HIV-Infected Patients Switched From a Protease Inhibitor Regimen (0518-033)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary efficacy analysis at Week 24 did not demonstrate non-inferiority of raltegravir versus lopinavir (+) ritonavir
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0518-033; 2007_508
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: HIV Infection
Keywords: treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Raltegravir & Placebo
  Interventions: Drug: Comparator: raltegravir; Drug: Comparator: placebo
- 2 (Active Comparator): Lopinavir (+) Ritonavir & Placebo
  Interventions: Drug: Comparator: lopinavir (+) ritonavir; Drug: Comparator: placebo

INTERVENTIONS:
Drug: Comparator: raltegravir — raltegravir 400 milligram (mg) by mouth (PO) twice daily (b.i.d) for up to 48 weeks of treatment
  Arms: 1
Drug: Comparator: placebo — lopinavir (+) ritonavir 400/100 mg by mouth (PO) twice daily (b.i.d.) Placebo for up to 48 weeks of treatment
  Arms: 1
Drug: Comparator: lopinavir (+) ritonavir — lopinavir (+) ritonavir 400/100 mg by mouth (PO) twice daily (b.i.d.) for up to 48 weeks of treatment
  Arms: 2
Drug: Comparator: placebo — raltegravir 400 mg by mouth (PO) twice daily (b.i.d.) Placebo for up to 48 weeks of treatment
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the efficacy, safety, and tolerability of an investigational treatment for patients with Human Immunodeficiency Virus (HIV).

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is human immunodeficiency virus (HIV) positive
* Patient has documented Human Immunodeficiency Virus (HIV) RiboNucleic Acid (RNA) <50 copies/milliliter (mL) for at least 3 months while on a KALETRA based regimen
* Patient has been on a KALETRA based regimen for at least 3 months without a change in background antiretroviral therapy
* Patient has no documentation of HIV RNA >50 copies/mL for at least 3 months while on the KALETRA based regimen

Exclusion Criteria:

* Patient is or plans to become pregnant, or is nursing a child
* Patient plans to donate eggs or impregnate/donate sperm
* Patient is receiving Stavudine (d4T) as a component of the background antiretroviral therapy
* Patient is currently receiving a second protease inhibitor in addition to KALETRA
* Patient is currently receiving, or has received in the past twelve weeks, treatment for the management of elevated lipids
* Patient has used another experimental HIV-integrase inhibitor
* Patient has a current (active) diagnosis of acute hepatitis due to any cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Eron JJ, Young B, Cooper DA, Youle M, Dejesus E, Andrade-Villanueva J, Workman C, Zajdenverg R, Fatkenheuer G, Berger DS, Kumar PN, Rodgers AJ, Shaughnessy MA, Walker ML, Barnard RJ, Miller MD, Dinubile MJ, Nguyen BY, Leavitt R, Xu X, Sklar P; SWITCHMRK 1 and 2 investigators. Switch to a raltegravir-based regimen versus continuation of a lopinavir-ritonavir-based regimen in stable HIV-infected patients with suppressed viraemia (SWITCHMRK 1 and 2): two multicentre, double-blind, randomised controlled trials. Lancet. 2010 Jan 30;375(9712):396-407. doi: 10.1016/S0140-6736(09)62041-9. Epub 2010 Jan 12. PMID 20074791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III; First Patient In: 11-Jun-2007; Last Patient Last Visit for Week 24 (primary endpoint): 17-Oct-
  2008
  34 Sites (US, Peru, Brazil, Colombia, Mexico, South Africa, Thailand, India, and Australia).
Pre-assignment Details: HIV-seropositive patients who were ≥18 years old, had documented HIV RNA <50 copies/mL for at least 3 months, had been on a KALETRA™-based regimen for at least 3 months without a change in background antiretroviral therapy, and had no documentation of HIV RNA >50 copies/mL for at least 3 months.
Groups:
- MK0518 400 mg b.i.d.: MK0518 400 mg, which can be taken by mouth (PO) twice a day (b.i.d.), approximately 12 hours (10 to 14 hours) apart without regard to food, and placebo to KALETRA™ , which can be taken by mouth (PO) twice a day (b.i.d.), approximately 12 hours (10 to 14 hours) apart without regard to food
- KALETRA™ 400/100 mg b.i.d.: KALETRA™ 400/100 mg, which can be taken by mouth (PO) twice a day (b.i.d.), approximately 12 hours (10 to 14 hours) apart without regard to food, and placebo to MK0518 , which can be taken by mouth (PO) twice a day (b.i.d.), approximately 12 hours (10 to 14 hours) apart without regard to food
Period: Overall Study
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Started | 176 | 179
Treated | 176 | 178
Completed | 166 | 172
Not Completed | 10 | 7
Not completed — Never Treated | 0 | 1
Not completed — Lack of Efficacy | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d. | Total
Number analyzed (Participants) | 176 | 178 | 354
Age, Continuous [Mean (Full Range); unit: Years] | 42.0 [21 to 71] | 41.9 [23 to 74] | 42.0 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 137 | 138 | 275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 73 | 141
  Not Hispanic or Latino | 108 | 105 | 213
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 26 | 28 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 33 | 25 | 58
  White | 85 | 81 | 166
  More than one race | 32 | 42 | 74
  Unknown or Not Reported | 0 | 0 | 0
Cluster of Differentiation 4 (CD4) Cell Count [Mean (Full Range); unit: cells/mm3] | 470.8 [16 to 1916] | 482.4 [100 to 1744] | 476.6 [16 to 1916]
Fasting (non-random) serum High-Density Lipoprotein-Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 46.5 (12.8) | 47.9 (12.7) | 47.2 (12.7)
Fasting (non-random) serum Low-Density Lipoprotein-Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 103.5 (41.0) | 104.3 (30.6) | 103.9 (36.2)
Fasting (non-random) serum cholesterol [Mean (Standard Deviation); unit: mg/dL] | 214.7 (69.7) | 210.8 (46.4) | 212.7 (59.2)
Fasting (non-random) serum triglyceride [Mean (Standard Deviation); unit: mg/dL] — Standard Deviation (Robust): calculated as interquartile range (IQR)/1.075, where IQR=3rd quartile-1st quartile.
  mg/dL | 204.5 (156.3) | 217.5 (156.3) | 212.5 (156.3)
Non-HDL-C [Mean (Standard Deviation); unit: mg/dL] | 168.2 (71.8) | 163.4 (45.7) | 165.8 (60.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Plasma Human Immunodeficiency Virus (HIV) RiboNucleic Acid (RNA) <50 Copies/mL at Week 24
Time Frame: 24 Weeks
Population: Full analysis set; one patient was excluded from the analysis because they did not have an HIV RNA test performed at Week 24 but had a test result of HIV RNA <50 copies/mL at Week 12 and Week 36.
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 175 | 178
Participants | 154 | 167

2. Primary Outcome: Number of Patients With Clinical Adverse Experiences (CAEs) Through 24 Weeks
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  With CAEs | 123 | 112
  Without CAEs | 53 | 66

3. Other Pre Specified Outcome: Number of Patients With Serious CAEs Through 24 Weeks
Description: Serious CAEs are any AEs occurring at any dose that; results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  With Serious CAEs | 4 | 8
  Without Serious CAEs | 172 | 170

4. Other Pre Specified Outcome: Number of Patients With Drug-related CAEs Through 24 Weeks
Description: Patients with drug-related (as assessed by an investigator who is a qualified physician, according to his/her best clinical judgement) CAEs.
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  With drug-related CAEs | 23 | 35
  Without drug-related CAEs | 153 | 143

5. Other Pre Specified Outcome: Number of Patients With Serious Drug-related CAEs Through 24 Weeks
Description: Serious CAEs are any AEs occurring at any dose that; results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose. Drug-related are as assessed by an investigator who is a qualified physician, according to his/her best clinical judgement
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  With Serious drugrelated CAEs | 0 | 0
  Without Serious drugrelated CAEs | 176 | 178

6. Other Pre Specified Outcome: Number of Patients That Died by 24 Week Last Patient Last Visit
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  Died | 0 | 0
  Did Not Die | 176 | 178

7. Other Pre Specified Outcome: Number of Patients That Discontinued Due to CAEs Through 24 Weeks
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  Discontinued with CAEs | 0 | 0
  Did Not Discontinue with CAEs | 176 | 178

8. Other Pre Specified Outcome: Number of Patients With Laboratory Adverse Experiences (LAEs) Through 24 Weeks
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  With LAEs | 8 | 6
  Without LAEs | 168 | 172

9. Other Pre Specified Outcome: Number of Patients With Drug-related LAEs Through 24 Weeks
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  With LAEs | 4 | 1
  Without LAEs | 172 | 177

10. Other Pre Specified Outcome: Number of Patients With Serious LAEs Through 24 Weeks
Description: Serious LAEs are any LAEs occurring at any dose that; results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  With LAEs | 0 | 0
  Without LAEs | 176 | 178

11. Other Pre Specified Outcome: Number of Patients That Discontinued Due to LAEs Through 24 Weeks
Time Frame: 24 Week last patient last visit
Population: All patients who took study medication were included in the analysis
Measure: Number; unit: Participants
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 176 | 178
Participants
  Discontinued with LAEs | 0 | 0
  Did Not Discontinue with LAEs | 176 | 178

12. Primary Outcome: Mean Percent Change From Baseline in Fasting Serum Cholesterol at Week 12
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 166 | 165
Percent Change | -12.41 (15.80) | 1.29 (15.81)

13. Primary Outcome: Mean Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 166 | 162
Percent Change | -14.77 (18.78) | 2.91 (20.26)

14. Primary Outcome: Mean Percent Change From Baseline in Fasting Serum Low-density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 161 | 162
Percent Change | 3.99 (33.11) | 0.55 (21.51)

15. Primary Outcome: Mean Percent Change From Baseline in Fasting Serum High-density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 166 | 162
Percent Change | -0.64 (20.14) | -2.50 (16.50)

16. Primary Outcome: Median Percent Change From Baseline in Serum Triglyceride at Week 12
Description: Standard Deviation (Robust): calculated as interquartile range (IQR)/1.075, where IQR=3rd quartile-1st quartile.
Time Frame: Baseline and Week 12
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Median (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 166 | 165
Percent Change | -42.82 (29.86) | 8.20 (52.73)

17. Secondary Outcome: Mean Percent Change From Baseline in Fasting Serum Cholesterol at Week 24
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 168 | 165
Percent Change | -13.64 (16.25) | 3.55 (15.50)

18. Secondary Outcome: Mean Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) at Week 24
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 168 | 162
Percent Change | -15.83 (19.88) | 5.26 (19.90)

19. Secondary Outcome: Mean Percent Change From Baseline in Fasting Serum Low-density Lipoprotein Cholesterol (LDL-C) at Week 24
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 163 | 162
Percent Change | 5.12 (35.65) | 6.06 (26.22)

20. Secondary Outcome: Mean Percent Change From Baseline in Fasting Serum High-density Lipoprotein Cholesterol (HDL-C) at Week 24
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 168 | 162
Percent Change | -1.77 (20.56) | -0.15 (16.62)

21. Secondary Outcome: Median Percent Change From Baseline in Serum Triglyceride at Week 24
Description: Standard Deviation (Robust): calculated as interquartile range (IQR)/1.075, where IQR=3rd quartile-1st quartile.
Time Frame: Baseline and Week 24
Population: Patients who had both baseline and at least one post-baseline measurement were included in the analysis
Measure: Median (Standard Deviation); unit: Percent Change
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Number analyzed (Participants) | 168 | 165
Percent Change | -44.50 (33.26) | 7.06 (55.42)

ADVERSE EVENTS:
Time Frame: Adverse experiences that occurred after randomization and through Week 24 last patient last visit (17-Oct-2008) were collected.
Arm/Group | MK0518 400 mg b.i.d. | KALETRA™ 400/100 mg b.i.d.
Serious Adverse Events (participants affected / at risk) | 4/176 | 8/178
Other Adverse Events (participants affected / at risk) | 94/176 | 84/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0518 400 mg b.i.d. (N=176) | KALETRA™ 400/100 mg b.i.d. (N=178)
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Appendicitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kaposi's sarcoma AIDS related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK0518 400 mg b.i.d. (N=176) | KALETRA™ 400/100 mg b.i.d. (N=178)
Abdominal distension (Gastrointestinal disorders) | 4 | 6
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 29
Dry mouth (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 2 | 6
Gastritis (Gastrointestinal disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 6 | 9
Vomiting (Gastrointestinal disorders) | 1 | 4
Fatigue (General disorders) | 5 | 6
Pyrexia (General disorders) | 5 | 5
Gastroenteritis (Infections and infestations) | 2 | 6
Genital herpes (Infections and infestations) | 4 | 2
Influenza (Infections and infestations) | 7 | 6
Nasopharyngitis (Infections and infestations) | 5 | 6
Pharyngitis (Infections and infestations) | 5 | 2
Respiratory tract infection (Infections and infestations) | 4 | 4
Sinusitis (Infections and infestations) | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 16 | 15
Alanine aminotransferase increased (Investigations) | 5 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Dizziness (Nervous system disorders) | 3 | 7
Headache (Nervous system disorders) | 13 | 7
Paraesthesia (Nervous system disorders) | 3 | 4
Depression (Psychiatric disorders) | 7 | 5
Insomnia (Psychiatric disorders) | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 5
Hypertension (Vascular disorders) | 5 | 2

LIMITATIONS AND CAVEATS:
Study was terminated after the primary efficacy analysis at Week 24 did not demonstrate non-inferiority of MK0518 versus KALETRA™.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.